CLINICAL TRIAL: NCT04481412
Title: The Role of Cetirizine in Androgenetic Alopecia in Females
Brief Title: Topical Cetirizine in Androgenetic Alopecia in Females
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Samar Farghali Farid, Head and professor of clinical pharmacy department, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Cetirizine in alopecia
Record Dates: First submitted 2020-07-15; First posted 2020-07-22 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Androgenetic Alopecia
Keywords: cetirizine; minoxidil; androgenetic alopecia (AGA); Female pattern hair loss (FPHL)
MeSH Terms: conditions — Alopecia | interventions — Cetirizine; Ethanol; Minoxidil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): (33) patients will apply topical minoxidil (5%) once daily and topical cetirizine (1%) once daily on their scalp for 6 months.
  Interventions: Drug: Topical cetirizine; Drug: Topical minoxidil
- Control group (Active Comparator): (33) patients will apply topical minoxidil (5%) once daily and placebo once daily on their scalp for 6 months.
  Interventions: Drug: Placebo; Drug: Topical minoxidil

INTERVENTIONS:
Drug: Topical cetirizine — Topical cetirizine 1% spray that will be prepared at Faculty of Pharmacy, Cairo University and will be applied once daily.
  Other Names: Cetirizine 1%
  Arms: Study group
Drug: Placebo — 96% ethanol that will be applied once daily.
  Other Names: 96% ethanol
  Arms: Control group
Drug: Topical minoxidil — Topical Minoxidil 5% that will be applied once daily.
  Other Names: Minoxidil 5%

SUMMARY:
Cetirizine is a safe and selective, second-generation histamine H1 receptor antagonist, widely used in daily practice. A study showed that cetirizine causes a significant reduction in both the inflammatory cell infiltrate and PGD2 production. A pilot study on topical cetirizine showed that cetirizine increased total hair density, terminal hair density and diameter. Also, its lower potential side effects if compared with other drugs commonly used for AGA, as minoxidil, can promote a wider use and better compliance of cetirizine in the future for the treatment of AGA. Combinations of therapies are likely to be more efficacious than single treatments.

Treatments to clinically improve scalp hair density and reduce mid-pattern thinning leading to improved scalp coverage are highly important for the affected women. On the basis of the above evidence and lacking studies that confirm the effectiveness of cetirizine in AGA treatment, the aim of this study is to evaluate the efficacy and tolerability of topical cetirizine in female patients with AGA.

DETAILED DESCRIPTION:
Androgenetic alopecia (AGA) is the most common form of alopecia in men and women. It is a hereditary, androgen-dependent, progressive thinning of scalp hair that follows a defined pattern. The disease mechanism is still relatively poorly understood, but involves a strong genetic contribution as well as some environmental input. AGA manifests as a noticeable reduction of scalp hair coverage, shorter miniaturized telogen vellus hair follicles, and significantly slower rates of hair growth. Approximately 6% to 38% of healthy women experience some degree of frontal and frontoparietal hair loss. AGA may have significant impact on quality of life in female patients. When female AGA is associated with high levels of androgens, systemic antiandrogenic therapy may be needed. However, treating it with oral antiandrogens is usually ineffective suggesting that most female AGA cases are not systemic androgen dependent and topical treatment may be more appropriate.

Currently, the only clinically validated and licensed medication approved for increasing hair density in women with AGA is 2 % minoxidil topical solution, and up to 5% minoxidil in several countries. The collective effects of minoxidil lead to increased cutaneous blood flow, prolongation of the anagen growth phase, and increase in the size of smaller hair follicles. However, it produces moderate results, and must continue to be used to have a continued benefit, and may produce adverse side effects. The use of higher concentrations of minoxidil in women is supported by results from an early study suggesting that concentrations higher than 2% could improve efficacy without increasing the rates of adverse events when applying not more than 60 mg of minoxidil per day.

Based on the hypertrichosis observed in patients treated with analogues of prostaglandin F2a (PGF2a) (i.e. latanoprost used for glaucoma), it was supposed that prostaglandins would have an important role in hair growth. Their action is variable depending on the class they belong to: prostaglandin E(PGE) and PGF2a play a generally positive role on the hair growth, while PGD2 has an inhibitory role on the hair growth. Elevated levels of prostaglandin D2 synthase (PGDS) were found at the messenger ribonucleic acid (mRNA) and protein levels in bald scalp versus haired scalp of men with AGA; as well as the enzymatic product of PGDS, (PGD2), is generally elevated in bald human scalp tissue.

Cetirizine is a safe and selective, second-generation histamine H1 receptor antagonist, widely used in daily practice. A study showed that cetirizine causes a significant reduction in both the inflammatory cell infiltrate and PGD2 production. However, these effects apparently are not related to its anti-H1 activity. A pilot study on topical cetirizine showed that cetirizine increased total hair density, terminal hair density and diameter. Also, its lower potential side effects if compared with other drugs commonly used for AGA, as minoxidil (which often cause of hypertrichosis, contact allergic dermatitis, headache and hypotension), can promote a wider use and better compliance of cetirizine in the future for the treatment of AGA. Combinations of therapies are likely to be more efficacious than single treatments.

Treatments to clinically improve scalp hair density and reduce mid-pattern thinning leading to improved scalp coverage are highly important for the affected women. On the basis of the above evidence and lacking studies that confirm the effectiveness of cetirizine in AGA treatment, the aim of this study is to evaluate the efficacy and tolerability of topical cetirizine in female patients with AGA.

ELIGIBILITY:
Inclusion Criteria:

1. Females with androgenetic alopecia of age 20-50 years.
2. Patients experiencing active hair loss within the last 12 months.
3. Sinclair scale 2, 3 and 4.
4. Patients willing to continue their current regimen of vitamins and nutritional supplements and not start any new vitamins or nutritional supplements for the duration of the study.
5. Patients willing to use a mild non-medicated shampoo and conditioner for the duration of the study.
6. Patients who did not receive topical or systemic treatment for androgenetic alopecia or prostaglandins in the last 6 months.

Exclusion Criteria:

* 1. Patients with a chronic dermatological condition (eczema, psoriasis, infection, etc) of the scalp other than FPHL.

  2. Subjects who had hair transplants, scalp reduction, current hair weave or tattooing in the target area, which makes it difficult to perform hair count assessment.

  3. Subjects who received radiation therapy to the scalp, or has had chemotherapy in the past year.

  4. Subjects who have a known underlying medical problem that could influence hair growth such as HIV infection, connective tissue disease, a thyroid condition, inflammatory bowel disease or other medical conditions, at the discretion of the investigator.

  5. Subjects with clinical diagnosis of alopecia areata or other non-AGA forms of alopecia.

  6. Pregnant or lactating females or planning to become pregnant for the duration of the study.

  7. Patients with severe cardiovascular disease, uncontrolled or untreated hypertension, arrythmia or clinically relevant hypotension.

  8. Subjects with hair loss for greater than 5 years, as medical therapy is unlikely to have much effect at restoring hair follicles inactive for that long of a period.

  9. The subject has known hypersensitivity or previous allergic reaction to any of the active or inactive components of the test articles.

  10. Patients using any medications that potentially cause drug-induced hair loss (e.g., depotestosterone, haloperidol, methotrexate, methylprednisolone, prednisone, testosterone, divalproex sodium) within the last 3 months.

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Females with androgenetic alopecia of age 20-50.
Enrollment: 66 (Actual)
Dates: Start 2020-07-25 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
The change from baseline in number of terminal hairs and vellus hair | baseline, 12, 24 weeks
  Trichoscopic evaluation: of frontal, occipital and temporal areas regarding the change from baseline in number of terminal hairs, growing hair and vellus hair.
The change from baseline in hair shaft thickness | baseline, 12, 24 weeks
  Trichoscopic evaluation: of frontal, occipital and temporal areas regarding the change from baseline in hair shaft thickness.
The change from baseline in terminal and vellus hair density | baseline, 12, 24 weeks
  Trichoscopic evaluation: of frontal, occipital and temporal areas regarding the change from baseline in number of follicular openings.
The change in patient self-assessment from baseline | baseline, 6, 12, 18, 24 weeks
  Patient self-assessment of hair growth will be determined by means of a set of predetermined 5 questions in Arabic, each of which asks the patient about a specific aspect of their hair compared with the start of the study.

SECONDARY OUTCOMES:
The change in hair growth from baseline using global photographic assessment | baseline, 12, 24 weeks
  Standardized photographs of the scalp will be taken.
  1. An expert panel of 3 blinded dermatologists will evaluate hair growth or loss from baseline by comparing baseline with follow-up photographs of each subject by means of a 7-point scale to answer the following question: "How would you subjectively rate the patient's hair growth at this time point compared to baseline?". The scale ranges from-3 ( greatly decreased) to +3 (greatly increased). Assessments will be made at the 12th and 24th week by comparing the global photographs taken at baseline with those taken at each visit.
  2. Investigator assessment: Same as the expert panel assessment.
Number of patients with adverse effects | 6, 12, 18, 24 weeks
  Reports of adverse effects or local intolerance, if any, will be collected at every visit.

CONTACTS AND LOCATIONS:
Overall Officials: Maggie Abbassi, PhD, Study Chair — Faculty of Pharmacy, Cairo University; Hanan Nada, PhD, Study Chair — Cairo University; Samar Farid, PhD, Principal Investigator — Faculty of Pharmacy, Cairo University
Locations (1):
- Al-Kasr Al-Ainy outpatient dermatology clinic, Cairo, ِAl-Kasr Al-Ainy, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jaworsky C, Kligman AM, Murphy GF. Characterization of inflammatory infiltrates in male pattern alopecia: implications for pathogenesis. Br J Dermatol. 1992 Sep;127(3):239-46. doi: 10.1111/j.1365-2133.1992.tb00121.x. PMID 1390168
- [Background] Guo H, Gao WV, Endo H, McElwee KJ. Experimental and early investigational drugs for androgenetic alopecia. Expert Opin Investig Drugs. 2017 Aug;26(8):917-932. doi: 10.1080/13543784.2017.1353598. Epub 2017 Jul 12. PMID 28689433
- [Background] Rossi A, Campo D, Fortuna MC, Garelli V, Pranteda G, De Vita G, Sorriso-Valvo L, Di Nunno D, Carlesimo M. A preliminary study on topical cetirizine in the therapeutic management of androgenetic alopecia. J Dermatolog Treat. 2018 Mar;29(2):149-151. doi: 10.1080/09546634.2017.1341610. Epub 2017 Jun 29. PMID 28604133
- [Derived] Bassiouny EA, El-Samanoudy SI, Abbassi MM, Nada HR, Farid SF. Comparison between topical cetirizine with minoxidil versus topical placebo with minoxidil in female androgenetic alopecia: a randomized, double-blind, placebo-controlled study. Arch Dermatol Res. 2023 Jul;315(5):1293-1304. doi: 10.1007/s00403-022-02512-2. Epub 2022 Dec 26. PMID 36571611